CLINICAL TRIAL: NCT01492764
Title: Ablation of Ventricular Fibrillation by Accurate Targeting of Arrhythmogenic Regions (AVATAR)
Acronym: AVATAR
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: AVATAR
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Ventricular Tachyarrhythmias
Keywords: Ventricular Tachyarrhythmia; Ablation; Electrophysiology; Human; Mapping
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Active Group: This group will receive brief ablation at localized sources (Focal Impulse and Rotor Modulation, FIRM)
- Control Group: This group receives traditional ablation for this disorder

SUMMARY:
This study will test the hypothesis that many human heart rhythm disorders are caused by small localized sources, where brief ablation may successfully eliminate the heart rhythm disorder.

DETAILED DESCRIPTION:
The investigators will enroll patients with documented rapid heart rates from the bottom chambers of the heart (ventricular tachyarrhythmias).

During electrophysiological study, the investigators will map the localized sources of these heart rhythm disorders.

1. The 'active' group will prospectively receive brief ablation at localized sources (Focal Impulse and Rotor Modulation, FIRM).
2. The control group will be a historical cohort who have received traditional ablation for this disorder.

All patients will be followed for up to 1 year to ensure that they have no recurrent arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

1. Documented ventricular tachyarrhythmias.
2. Undergoing clinically indicated EP study with ablation.

Exclusion Criteria:

1. Unwillingness or inability to provide informed consent.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with documented rapid heart rhythms involving the bottom chambers of the heart.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
reduction in ventricular tachyarrhythmias events | 3 months
  Using careful clinical monitoring, we will compare the burden of VT/VF after ablation (including FIRM) to the burden preceding ablation.
safety of ventricular basket mapping in patients undergoing ablation | 1 month
  To assess the incidence of adverse events arising from ablation using basket mapping in the ventricles. These include but are not limited to stroke, systemic thromboembolism, MI or acute coronary syndrome, groin complications, or death.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Narayan, MD, PhD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California, San Diego Medical Center, San Diego, California
  - Veterans Affairs San Diego Medical Center, San Diego, California